CLINICAL TRIAL: NCT05246150
Title: The Effect Of Nursıng Practıces On The Near Infrared Spectroscopy Levels Of Premature Infants
Brief Title: NIRS Levels of Infants in Neonatal Intensive Care
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ezgi Ayvaz, NURSE, Eskisehir Osmangazi University
Other Study IDs: EsksehirOU
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infants receiving nursing care
  Interventions: Behavioral: nursing care practices

INTERVENTIONS:
Behavioral: nursing care practices — To determine the effect of nursing care practices on Near Infrared Spectroscopy (NIRS) levels in premature babies

SUMMARY:
Aim: This study was conducted to determine the effect of nursing care practices on the Near Infrared Spectroscopy (NIRS) levels of premature infants in the neonatal intensive care unit (NICU).

Materials and Method: This is a cross-sectional, analytical study. It was conducted over the period March 1 - April 26, 2019 in the Neonatal Intensive Care Unit (NICU) of Eskişehir Osmangazi University (ESOGU) Health Practices and Research Hospital. We did not calculate sample size, but included in the study, after the parents had been informed about the research, the entire universe of neonates in the NICU who matched the inclusion criteria during the period March 1 - April 26, 2019. The study was completed with 40 neonates. Data collection was performed with a "Descriptive Data Form," and a "Procedures Performed Chart." The data were evaluated with the IBM SPSS 24 package program.

ELIGIBILITY:
Inclusion Criteria:

* Neonates younger than a gestational age of 37 weeks
* Those monitored in an open or closed incubator

Exclusion Criteria:

* Intubated neonates connected to a mechanical ventilator
* Infants of a gestational age of 37 weeks or more
* Infants under sedation
* Infants with neurological illness (e.g., hypoxic ischemic encephalopathy, hydrocdphalus)

Ages: 1 Day to 40 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 40 premature newborns
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
nursing practices | 24 hours
  Change of nursing practices on Near Infrared Spectroscopy levels

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided